CLINICAL TRIAL: NCT07066345
Title: Comparing Integrative Interventions for Chronic Pelvic Pain
Acronym: CII-CPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Till, MD, MPH (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Sara Till, MD, MPH, Assistant Professor of Obstetrics and Gynecology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00273882; K23HD099283 (NIH)
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Pain
Keywords: Chronic pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Patients will be blinded to their group assignment. Study team members involved in outcome assessment will be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1- My Pelvic Plan (Experimental): Patients will be randomized to receive one of two non-pharmacologic interventions. Group 1 will receive access to a novel web-based, cognitive behavioral program.
  Interventions: Device: My Pelvic Plan
- Group 2- Bend (Active Comparator): Patients will be randomized to receive one of two non-pharmacologic interventions. Group 2 will receive a subscription to a commercially available remote application.
  Interventions: Behavioral: Bend

INTERVENTIONS:
Device: My Pelvic Plan — My Pelvic Plan is comprised of a self-guided program that combines education on several individual conditions that often contribute to CPP, and will include instruction on cognitive and behavioral restructuring techniques that can help to manage chronic pelvic pain symptoms.
  Arms: Group 1- My Pelvic Plan
Behavioral: Bend — Bend is a highly rated physical activity application that helps guide users through gentle stretching and yoga poses.
  Arms: Group 2- Bend

SUMMARY:
The researchers will conduct a pilot randomized trial to assess functional changes with two different remote integrative non-pharmacologic interventions for women with chronic pelvic pain (CPP). The study team will compare a novel web-based, cognitive-behavioral program designed for patients with CPP and a commercially available physical activity remote application. The team aims to gather information about differences in sexual function, physical function, pain, and quality of life.

DETAILED DESCRIPTION:
My Pelvic Plan was determined as a medical device under FDA enforcement discretion.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a new patient visit with the Chronic Pelvic Pain and Endometriosis Referral Clinic within the Department of Obstetrics and Gynecology at the University of Michigan for treatment of chronic pelvic pain.
* Have chronic pelvic pain, defined as moderate to severe pelvic pain that is ≥ 4 on a 0-10 numeric rating scale (worst pain during the day) for ≥ 6-month duration, and is non-cyclic, occurring for at least 14 days of each month.
* Report moderate to severe sexual dysfunction or sexual restriction on CPP clinic intake questionnaire. This will be defined as the patient indicating one of the following responses to a question that asks them to describe their experience relative to sexual activity: my sex life is nearly normal but is very painful, my sex life is severely restricted by pain, my sex life is nearly absent because of pain, pain prevents any self life at all.
* Have access to internet via computer and must have a smartphone
* Willing to download and use the Bend application on their smartphone if they are randomized to that intervention
* English-language proficiency (current version of the My Pelvic Plan website is in English)

Exclusion Criteria:

* Pregnancy (at time of screening visit). Participants will be allowed to continue to study if they become pregnant during the study period.
* Severe physical impairment precluding participating in internet-based program or remote application (for example, complete blindness or deafness)
* Medical condition that precludes low-intensity, short-duration physical activity and gentle stretching, including cerebral palsy, severe hip or knee osteoarthritis, severe heart failure, severe Chronic obstructive pulmonary disease (COPD) requiring oxygen use
* Prior care within the Chronic Pelvic Pain and Endometriosis Referral Clinic within the Department of Obstetrics and Gynecology at the University of Michigan for treatment of chronic pelvic pain (seen previously but meets criteria for new patient visit because > 3 year interval since last clinic visit).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-01-19 (Actual); Study Completion 2026-01-19 (Actual)

PRIMARY OUTCOMES:
Total score on the Female Sexual Function Index (FSFI) | 8 weeks
  This female sexual function index (FSFI) questionnaire calculator evaluates and monitors woman sexual functioning as well as the level of dysfunction. The FSFI ranges in scores from 2-36 where higher scores indicate more disfunction. (0's may indicate no sexual activity in period in question.)
PROMIS-29 Profile v2.1 physical function domain score | 8 weeks
  PROMIS-29 Profile v2.1 is a questionnaire covering 7 domains including physical function. Higher scores indicate more severity/worse health.
PROMIS-29 Profile v2.1 pain interference domain score | 8 weeks
  PROMIS-29 Profile v2.1 is a questionnaire covering 7 domains including pain interference. Higher scores indicate more severity/worse health.

SECONDARY OUTCOMES:
Total score on the Female Sexual Function Index (FSFI) | 4 weeks
  This female sexual function index (FSFI) questionnaire calculator evaluates and monitors woman sexual functioning as well as the level of dysfunction. The FSFI ranges in scores from 2-36 where higher scores indicate more disfunction. (0's may indicate no sexual activity in period in question.)
PROMIS-29 Profile v2.1 pain interference domain score | 4 weeks
  PROMIS-29 Profile v2.1 is a questionnaire covering 7 domains including pain interference. Higher scores indicate more severity/worse health.
PROMIS-29 Profile v2.1 physical function domain score | 4 weeks
  PROMIS-29 Profile v2.1 is a questionnaire covering 7 domains including physical function. Higher scores indicate more severity/worse health.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Till, MD MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT07066345/ICF_000.pdf